CLINICAL TRIAL: NCT01374087
Title: Proof-of-concept Multicentre, Prospective, Randomised, Open-label- Parallel-group Clinical Trial to Assess the Efficacy of Brachytherapy With or Without Hormone Therapy Using Triptorelin 22.5 mg 6-month Formulation in Patients With Recurrence of Prostate Cancer Previously Treated With Radiotherapy
Brief Title: Study to Assess the Efficacy of Brachytherapy With or Without Hormone Therapy, Using Triptorelin 22.5mg in Patients With Recurrence of Prostate Cancer
Acronym: ANABRAQ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment of patients.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-92-52014-177; 2010-019158-41 (EudraCT Number)
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: Recurrent Prostate Carcinoma; Brachytherapy; Triptorelin; Hormone Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brachytherapy + Triptorelin 22.5 mg (Experimental): Brachytherapy: Low or high dose rate. Triptorelin: A single, intramuscular injection (22.5 mg), preferably 2 months before brachytherapy.
  Interventions: Drug: Triptorelin 22.5 mg; Radiation: Brachytherapy
- Brachytherapy (Active Comparator): Brachytherapy: Low or high dose rate.
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Drug: Triptorelin 22.5 mg — Triptorelin: A single, intramuscular injection (22.5 mg), preferably 2 months before brachytherapy.
  Arms: Brachytherapy + Triptorelin 22.5 mg
Radiation: Brachytherapy — Brachytherapy: Low or high dose rate.

SUMMARY:
The primary objective of the study was to compare the efficacy of brachytherapy versus brachytherapy + triptorelin 22.5 mg (single injection) in subjects with recurrence of prostate cancer previously treated with radiotherapy. Efficacy was to be assessed by biochemical failure-free survival (BFFS) curves from treatment initiation up to 5 years.

Secondary objectives included comparing the following: the differences in time to progression of subjects receiving brachytherapy + triptorelin 22.5 mg versus subjects receiving brachytherapy only, the BFFS percentages between both treatment groups at 5 years from treatment initiation, overall survival between both treatment groups, total testosterone changes (from baseline visit up to 12 months) and Prostate Specific Antigen (PSA) levels (from baseline visit up to 60 months of treatment) between both treatment groups, quality of life (QoL) modifications (Spanish version of the Expanded Prostate Cancer Index Composite (EPIC) questionnaire) between the baseline score and the rest of measurements, and to compare safety between both treatment groups.

DETAILED DESCRIPTION:
This was a proof-of-concept, prospective, parallel, multicentre, randomised and open-label trial, including a follow-up of all subjects conducted at 11 centres in Spain. Study visits included an inclusion visit (Visit 1), a treatment administration visit (Visit 2), and 9 follow-up visits (Visit 3 to Visit 11) from 3 to 60 months after study treatment administration. All of the procedures performed at these visits were in accordance with routine clinical practice. Subjects were randomised to any one of the two treatment arms (Group 1: brachytherapy only, or Group 2: brachytherapy + triptorelin 22.5 mg). Randomisation was stratified according to the brachytherapy dose rate (low or high dose rate).

Visit 1 included the collection of demographic data, a review of clinical details of prostate cancer and its treatment, blood sampling (for Prostate Specific Antigen (PSA), testosterone, and haematology and biochemistry parameters, as appropriate), administration of the QoL questionnaire and International Prostatic Symptom Score (IPSS), and treatment group allocation. Visit 2 included a review of the eligibility criteria, recording of concomitant medications and adverse events (AEs) and study drug administration. Visits 3 to 11 included recording of AEs and concomitant medications, blood sampling and administration of the QoL questionnaire and IPSS.

Following the selection visit (Visit 1), all subjects were scheduled to brachytherapy. Those subjects who were randomised to the concomitant hormone therapy group received a single dose of triptorelin 22.5 mg by intramuscular injection at Visit 2, 2 weeks following the selection visit (Visit 1), and preferably 2 months before receiving brachytherapy. One week before and two weeks after triptorelin administration, subjects were permitted to receive an anti-androgen to counteract a transient increase in testosterone levels.

The study was prematurely stopped due to the slow enrolment of subjects. Of the planned 86 evaluable subjects, 35 were screened, and 32 were randomised between 3 November 2011 and 26 May 2014. The slow inclusion of subjects was due to several factors, among which there were changes in clinical practice which caused such subjects to be offered alternative treatments to brachytherapy. Due to the small number of subjects, none of the planned efficacy analyses were performed. Instead, the data were analysed as follows:

* Efficacy data and quality of life (QoL) outcomes were displayed only in listings.
* Safety information was displayed using listings and summary tables.

ELIGIBILITY:
Inclusion Criteria:

1. A history of prostate cancer (T1-T2-T3 N0 M0), confirmed through histopathology and initially treated with radiotherapy.
2. Age ≤ 75 years.
3. Biochemical failure due to Phoenix criteria (nadir + 2) and local recurrence of the initial prostate cancer, confirmed by prostate biopsy, with neither regional involvement nor distant metastases.
4. Late local recurrence of the initial prostate cancer. A recurrence is late when it appears after longer than 18 months post-radiotherapy.
5. PSA < 10 ng/mL at the time of recurrence.
6. The subject was required to be amenable to brachytherapy treatment.
7. Adequate urinary function according to the questionnaire (IPSS ≤ 20 points).
8. Suitable bone marrow function, determined by:

   * Haemoglobin > 10 g/dL.
   * Neutrophil count > 1.5 x 10^9/L.
   * Platelet count > 100 x 10^9/L.
9. Suitable liver function determined by: serum bilirubin < 1.5 x Upper Normal Level (UNL), and alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5xUNL.
10. Suitable renal function determined by: serum creatinine < 1.5 x UNL, or creatinine clearance ≥ 60 mL/min.
11. The subject was required to be ≥ 18 years old.
12. The subject had to give his written informed consent (personally signed and dated) before starting with any study-related procedure.
13. Life expectancy > 5 years.

Exclusion Criteria:

1. Evidence of metastatic disease.
2. Previous evidence of hormone-resistant cancer.
3. Lack of availability for performing regular follow-up.
4. Subjects who were receiving or had received either luteinizing hormone-releasing hormone (LH-RH) agonists, or antagonists, over the previous 12 months.
5. Subjects who had been on treatment with other hormone therapies, including antagonists, megestrol acetate, finasteride, dutasteride, any herbaceous product known to reduce the PSA levels, or any systemic corticosteroid, over the previous 4 weeks.
6. Subjects who had previously undergone a radiotherapy treatment that was completed within 18 months of inclusion.
7. Subjects with pre-existing heart failure (New York Heart Association class III or IV), or with a myocardial infarction within 6 months of inclusion.
8. Subjects with a significant co-existing disease or an active infection.
9. Subjects who had been treated with investigational therapies within 4 weeks prior to the brachytherapy ± triptorelin treatment.
10. Subjects with known hypersensitivity to triptorelin, LH-RH, other LH-RH-analogous agonists, or any excipients in triptorelin 22.5 mg.
11. Subjects with a mental condition that prevented them from understanding the nature, the scope and the potential consequences of this study, and/or subjects who showed an uncooperative attitude.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (11):
- Spain (11):
  - Fundación IMOR, Barcelona
  - H. de la Santa Creu i Sant Pau, Barcelona
  - ICO Institut Català d'Oncologia-Hospitalet, L'Hospitalet de Llobregat
  - H. Ramón y Cajal, Madrid
  - H. Sanchinarro, Madrid
  - H. Carlos Haya, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Instituto Oncológico, San Sebastián
  - H. Universitario Marqués de Valdecilla, Santander
  - IVO Instituto Valenciano de Oncología, Valencia
  - H. Do Meixoeiro, Vigo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with recurrence of prostate cancer previously treated with radiotherapy were recruited in 11 sites in Spain from November 2011 until December 2014 when the study was prematurely discontinued.
Pre-assignment Details: 35 subjects were screened and 3 did not meet inclusion criteria. Of those who met the inclusion criteria and none of the exclusion criteria, 32 were randomised to treatment and 31 received treatment after 1 subject (in the Brachytherapy + Triptorelin arm) withdrew consent.
Groups:
- Brachytherapy: Subjects were randomised to receive brachytherapy alone, as either a low dose rate ([125]I) or high dose rate ([192]I).
- Brachytherapy + Triptorelin 22.5 mg: Subjects received brachytherapy as either a low dose rate ([125]I) or high dose rate ([192]I). Subjects also received a single intramuscular injection of 22.5 milligrams (mg) triptorelin at Visit 2 (Day 1).
Period: Overall Study
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Started (Subjects treated) | 16 | 15
Completed | 0 | 0
Not Completed | 16 | 15
Not completed — Adverse Event | 1 | 0
Not completed — Disease progression | 2 | 2
Not completed — Study discontinued | 13 | 13

BASELINE CHARACTERISTICS:
Population: Safety population: Safety population consisted of all randomised subjects who received at least one dose of study medication. Subjects were allocated to the treatment they actually received.
Groups:
- Brachytherapy + Triptorelin 22.5 mg: Subjects received brachytherapy as either a low dose rate ([125]I) or high dose rate ([192]I). Subjects also received a single intramuscular injection of 22.5 mg triptorelin at Visit 2 (Day 1).
- Total: Total of all reporting groups
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Median (Full Range); unit: years] | 67.50 [59.0 to 76.0] | 70.00 [58.0 to 76.0] | 68.00 [58.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 15 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 16 | 15 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Failure-free Survival (BFFS)
Description: BFFS was determined by a prostate-specific antigen (PSA) increase of 2 nanograms per millilitre (ng/mL) or more in comparison with the pre-study nadir PSA and confirmed in the course of follow-up by a second value 3 weeks later or longer over the 5 year follow-up. Time to BFFS was defined from treatment initiation to the first time when PSA increase of 2 ng/mL was observed.
  As the study was prematurely terminated, no analyses were conducted. Data for BFFS are listed by subject for those individuals who reported biochemical failure. Time (in months) to biochemical failure is relative to the date of brachytherapy.
Time Frame: Up to 5 years
Population: A total of 3 subjects in each treatment group reported biochemical failure. The subject numbers assigned in the study are not presented. The subjects with biochemical failure are listed as Subject 1 to Subject 6, with these bearing no relation to the subject numbers used for other endpoints herein.
Measure: Number; unit: Months
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Number analyzed (Participants) | 3 | 3
Months
  Subject 1 | 5.2 | NA — Subject not treated in this study arm.
  Subject 2 | 12.2 | NA — Subject not treated in this study arm.
  Subject 3 | 5.7 | NA — Subject not treated in this study arm.
  Subject 4 | NA — Subject not treated in this study arm. | 24.7
  Subject 5 | NA — Subject not treated in this study arm. | 29.9
  Subject 6 | NA — Subject not treated in this study arm. | 5.6

2. Secondary Outcome: Time to Progression
Description: Time to progression (in months) was measured from the informed consent date to the date of first event occurrence. Progression was defined as either: death from all causes or disease progression (defined as PSA increased by 2 ng/mL as compared to the pre-trial nadir PSA, confirmed during follow-up by a second value after 3 or more weeks, or the diagnosis of a new clinical recurrence of their prostate cancer (metastasis, new injury, etc.)).
  As the study was prematurely terminated, no analyses were conducted. Data for time to progression are listed by subject for those individuals who reported progression.
Time Frame: Up to 5 years
Population: A total of 3 subjects in the brachytherapy group and 4 subjects in the brachytherapy + triptorelin 22.5 mg group reported treatment failure. The subject numbers assigned in the study are not presented. The subjects with progression are listed as Subjects 1 to 7, with these bearing no relation to the subject numbers used for other endpoints herein.
Measure: Number; unit: Months
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Number analyzed (Participants) | 3 | 4
Months
  Subject 1 | 6.7 | NA — Subject not treated in this study arm.
  Subject 2 | 12.6 | NA — Subject not treated in this study arm.
  Subject 3 | 6.5 | NA — Subject not treated in this study arm.
  Subject 4 | NA — Subject not treated in this study arm. | 27.2
  Subject 5 | NA — Subject not treated in this study arm. | 30.8
  Subject 6 | NA — Subject not treated in this study arm. | 16.8
  Subject 7 | NA — Subject not treated in this study arm. | 12.8

3. Secondary Outcome: BFFS Percentage 5 Years From Treatment Initiation
Description: A subject had a biochemical failure if there was an increase of PSA of 2 ng/mL or more in comparison with the pre-study nadir PSA confirmed in the course of follow-up by a second value after 3 or more weeks or with diagnosis of a new clinical recurrence of their prostate cancer over the 5 year follow-up.
Time Frame: 5 years
Population: No data analyses were conducted as the study was terminated prior to completion of the 5-year follow-up.
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months from diagnosis (biopsy date for local recurrence) to death due to any cause, the last visit or the loss to follow-up.
Time Frame: 5 years
Population: No data analyses for Overall Survival were conducted as the study was terminated prior to completion of the 5 year follow-up.
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Change in Total Serum Testosterone Levels From Baseline at 3, 6 and 12 Months
Description: Blood samples were drawn for serum testosterone at baseline (Visit 1) and then at 3, 6 and 12 months.
  Changes from baseline in total serum testosterone levels in relation to the normal parameter ranges are indicated. WNR = Within Normal Range, BNR= Below Normal Range and ANR = Above Normal Range.
Time Frame: Baseline and 3, 6 and 12 months
Population: The Safety population consisted of all randomised subjects who received at least one dose of study medication. Only subjects with data available at each timepoint are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Number analyzed (Participants) | 16 | 15
Participants
  WNR at Baseline and Month 3: number analyzed (Participants) | 7 | 9
  WNR at Baseline and Month 3 | 6 | 0
  WNR at Baseline, BNR at Month 3: number analyzed (Participants) | 7 | 9
  WNR at Baseline, BNR at Month 3 | 1 | 7
  BNR at Baseline and Month 3: number analyzed (Participants) | 7 | 9
  BNR at Baseline and Month 3 | 0 | 2
  WNR at Baseline and Month 6: number analyzed (Participants) | 6 | 9
  WNR at Baseline and Month 6 | 5 | 2
  WNR at Baseline, BNR at Month 6: number analyzed (Participants) | 6 | 9
  WNR at Baseline, BNR at Month 6 | 1 | 5
  BNR at Baseline and Month 6: number analyzed (Participants) | 6 | 9
  BNR at Baseline and Month 6 | 0 | 2
  WNR at Baseline and Month 12: number analyzed (Participants) | 6 | 7
  WNR at Baseline and Month 12 | 3 | 4
  WNR at Baseline, BNR at Month 12: number analyzed (Participants) | 6 | 7
  WNR at Baseline, BNR at Month 12 | 3 | 2
  BNR at Baseline and Month 12: number analyzed (Participants) | 6 | 7
  BNR at Baseline and Month 12 | 0 | 1

6. Secondary Outcome: Number of Participants With Change in Total Serum PSA Levels From Baseline at 3, 6 and 12 Months
Description: Blood samples were drawn for serum PSA at baseline (Visit 1) and at 3, 6 and 12 months.
  Changes from baseline in total serum PSA levels in relation to the normal parameter ranges are indicated. WNR = Within Normal Range, BNR= Below Normal Range and ANR = Above Normal Range.
Time Frame: Baseline and 3, 6 and 12 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Number analyzed (Participants) | 16 | 15
Participants
  WNR at Baseline and Month 3: number analyzed (Participants) | 12 | 7
  WNR at Baseline and Month 3 | 3 | 2
  ANR at Baseline and Month 3: number analyzed (Participants) | 12 | 7
  ANR at Baseline and Month 3 | 2 | 0
  ANR at Baseline, WNR at Month 3: number analyzed (Participants) | 12 | 7
  ANR at Baseline, WNR at Month 3 | 7 | 5
  WNR at Baseline and Month 6: number analyzed (Participants) | 11 | 9
  WNR at Baseline and Month 6 | 2 | 5
  WNR at Baseline, BNR at Month 6: number analyzed (Participants) | 11 | 9
  WNR at Baseline, BNR at Month 6 | 0 | 1
  ANR at Baseline and Month 6: number analyzed (Participants) | 11 | 9
  ANR at Baseline and Month 6 | 3 | 0
  ANR at Baseline and WNR at Month 6: number analyzed (Participants) | 11 | 9
  ANR at Baseline and WNR at Month 6 | 6 | 3
  WNR at Baseline and Month 12: number analyzed (Participants) | 6 | 8
  WNR at Baseline and Month 12 | 1 | 4
  WNR at Baseline, BNR at Month 12: number analyzed (Participants) | 6 | 8
  WNR at Baseline, BNR at Month 12 | 0 | 1
  ANR at Baseline and Month 12: number analyzed (Participants) | 6 | 8
  ANR at Baseline and Month 12 | 1 | 0
  ANR at Baseline, WNR at Month 12: number analyzed (Participants) | 6 | 8
  ANR at Baseline, WNR at Month 12 | 4 | 3

7. Secondary Outcome: Change in Quality of Life (QoL) Modifications (Spanish Version of the Expanded Prostate Cancer Index Composite (EPIC) Questionnaire) From Baseline at 5 Years
Description: EPIC assessed the disease-specific aspects of prostate cancer and its therapies and comprised four summary domains (Urinary, Bowel, Sexual and Hormonal). Factor analysis supported dividing the Urinary Domain Summary Score into two different Incontinence and Irritative/Obstructive subscales. In addition, each Domain Summary Score had measurable Function Subscale and Bother Subscale components. Response options for each EPIC item formed a Likert scale, and multi-item scale scores were transformed linearly to a 0-100 scale, with higher scores representing better Health-Related QoL.
Time Frame: Baseline and 5 years.
Population: No data analyses for change from baseline score for QoL modifications were conducted as the study was terminated prior to completion of the 5 year follow-up.
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from treatment initiation (Day 1) to end of the study (up to 5 years).
Description: The Safety population consisted of all randomised subjects who received at least 1 dose of study medication.
Arm/Group | Brachytherapy | Brachytherapy + Triptorelin 22.5 mg
Serious Adverse Events (participants affected / at risk) | 3/16 | 2/15
Other Adverse Events (participants affected / at risk) | 11/16 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brachytherapy (N=16) | Brachytherapy + Triptorelin 22.5 mg (N=15)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brachytherapy (N=16) | Brachytherapy + Triptorelin 22.5 mg (N=15)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 1 (1) | 0 (0)
Erythrasma (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (4) | 4 (5)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Hypertonic bladder (Renal and urinary disorders) | 2 (3) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (2)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely stopped due to slow enrolment and all subjects were withdrawn following study termination in December 2014. Due to the small number of participating subjects very limited analyses were performed for the efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor required reasonable opportunity to review any summary, presentation, or paper before the material was submitted for publication or communicated. This also applied to any amendments that were requested by evaluators or journal directors. The Sponsor committed to comment on the draft documents within a time period agreed in the contractual provisions between the Sponsor and authors or their institutions. Delays were also possible if publication would adversely affect patentability.